CLINICAL TRIAL: NCT03839602
Title: Delineation of Reducing Clinical Target Volume for Early-stage Nasopharyngeal
Brief Title: Delineation of Reducing Clinical Target Volume for Early-stage Nasopharyngeal Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTV Delineation in I-II NPC
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Target Volume Delineation; Early-stage Nasopharyngeal Carcinoma; Intensity Modulated Radiation Therapy
Keywords: Locoregional Failure Pattern; Toxicity
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Intervention Model Description: The CTV was divided into CTV1 (high risk) and CTV2 (low risk) according to the biological behavior and characteristics of early-stage NPC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- reducing CTV (Experimental): The gross tumor volume of the nasopharynx and neck nodes (GTVnx and GTVnd) were delineated according to the tumor extension. The CTV was divided into CTV1 (high risk) and CTV2 (low risk) according to the biological behavior and characteristics of early-stage NPC. The prescribe doses of GTVnx, GTVnd, CTV1 and CTV2 were 68Gy, 60-66Gy, 60Gy and 50-54Gy in 30 fractions, respectively.
  Interventions: Radiation: Reducing CTV

INTERVENTIONS:
Radiation: Reducing CTV — CTVs were delineated in line with tumor stage, i.e. tumor invasion.

SUMMARY:
To analyze the long-term results and toxicities of the reducing clinical target volume (CTV) delineation method in early-stage nasopharyngeal carcinoma (NPC) patients treated with intensity modulated radiation therapy (IMRT).

DETAILED DESCRIPTION:
The investigators designed a prospective phase II study for early-stage NPC patients, and proposed a reasonable delineation method of reducing CTV according to the clinical characteristics and tumor infiltration patterns, performing therapeutic dose to tumor and prophylactic dose to CTV while protecting as much normal tissues as possible, in order to ensure a long-term survival with good quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed NPC (WHO II-III)
2. stage I-IIb according to the 6th AJCC/UICC
3. no previous treatment for NPC
4. between 18 and 70 years old
5. KPS ≥ 80 scores
6. adequate organ function (white blood cell ≥ 4.0×109/L; absolute neutrophil count ≥ 1.5×109/L; hemoglobin ≥ 100g/L; platelet count ≥ 100×109/L; total bilirubin, aspartate aminotransferase and alanine aminotransferase ≤ 1.5X upper limit normal; and creatinine clearance rate ≥ 30 mL/min)

Exclusion Criteria:

1. fine-needle aspiration biopsy, incisional or excisional biopsy of neck lymph node, or neck dissection prior IMRT
2. disease progression during IMRT
3. presence of distant metastasis
4. pregnancy or lactation
5. previous malignancy or other concomitant malignant disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2001-05-01 (Actual); Primary Completion 2006-10-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
LRRFS | 5 year
  locoregional recurrence free survival

SECONDARY OUTCOMES:
Locoregional failure patterns | 5 year
  To identify the locoregional failure patterns: in-field recurrence, marginal recurrence and out-field recurrence
DMFS | 5 year
  distant metastasis free survival
DSS | 5 year
  disease specific survival
OS | 5 year
  overall survival
Acute toxicity assessed with National Cancer Institute Common Toxicity Criteria for Adverse Events version 3.0 (NCI-CTCAE v3.0) | 3 months after IMRT
  National Cancer Institute Common Toxicity Criteria for Adverse Events version 3.0 (NCI-CTCAE v3.0)
Late toxicity assessed with Radiation Therapy Oncology Group radiation morbidity scoring criteria | 5 year
  Radiation Therapy Oncology Group radiation morbidity scoring criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Miao J, Di M, Chen B, Wang L, Cao Y, Xiao W, Wong KH, Huang L, Zhu M, Huang H, Huang S, Han F, Deng X, Xiang Y, Lv X, Xia W, Tan SH, Wee JTS, Guo X, Chua MLK, Zhao C. A Prospective 10-Year Observational Study of Reduction of Radiation Therapy Clinical Target Volume and Dose in Early-Stage Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):672-682. doi: 10.1016/j.ijrobp.2020.03.029. Epub 2020 Apr 6. PMID 32272183